CLINICAL TRIAL: NCT03395002
Title: Comparison of Bronchodilator Efficacy of Tiotropium/Salmeterol/Fluticasone 9/50/500 mcg Combination Treatment Administered Via Discair® With Original Products Seretide Diskus 500 mcg Inhalation Powder Plus Spiriva 18 mcg Inhalation Powder Treatment in Patients With Moderate-severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Tiotropium/Salmeterol/Fluticasone Fixed Dose Combination Tratment Via Discair vs Tiotropium Via Handihaler + Salmeterol/Fluticasone Via Diskus Free Combination Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEU-01.17
Record Dates: First submitted 2017-12-07; First posted 2018-01-09 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2019-01

CONDITIONS: COPD
Keywords: Tiotropium; Salmeterol; Fluticasone; COPD; Bronchodilator effect; Discair; Diskus; Spirometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tiotropium/Salmeterol/Fluticasone (Experimental): Tiotropium/Salmeterol/Fluticasone 9/50/500 mcg Inhalation Powder (1 puff) twice daily (approximately every 12 hr) via Discair®
  Interventions: Drug: Tiotropium/Salmeterol/Fluticasone 9/50/500 mcg Inhalation Powder
- Tiotropium + Salmeterol/Fluticasone (Active Comparator): Tiotropium 18 mcg Inhalation Powder (1 puff) once daily via Handihaler® + Salmeterol/Fluticasone 50/500 mcg Inhalation Powder (1 puff) twice daily (approximately every 12 hr) via Diskus®
  Interventions: Drug: Tiotropium 18 mcg Inhalation Powder; Drug: Salmeterol/Fluticasone 50/500 mcg Inhalation Powder

INTERVENTIONS:
Drug: Tiotropium/Salmeterol/Fluticasone 9/50/500 mcg Inhalation Powder — Tiotropium/Salmeterol/Fluticasone 9/50/500 mcg Inhalation Powder (1 puff) twice daily via Discair® for two days.
  Other Names: Saltif 9/50/500 mcg Inhalation Powder
  Arms: Tiotropium/Salmeterol/Fluticasone
Drug: Tiotropium 18 mcg Inhalation Powder — Tiotropium 18 mcg Inhalation Powder (1 puff) once daily via Handihaler® for two days.
  Other Names: Spiriva 18 mcg Inhalation Powder
  Arms: Tiotropium + Salmeterol/Fluticasone
Drug: Salmeterol/Fluticasone 50/500 mcg Inhalation Powder — Salmeterol/Fluticasone 50/500 mcg Inhalation Powder (1 puff) twice daily (approximately every 12 hr) via Diskus® for two days
  Other Names: Seretide Diskus® 500 mcg Inhalation Powder
  Arms: Tiotropium + Salmeterol/Fluticasone

SUMMARY:
The overall objective is to asses the bronchodilator effect of Tiotropium/Salmeterol/Fluticasone combination delivered via Discair® twice daily as compared with original products Seretide Diskus 500 mcg Inhalation Powder twice daily and Spiriva 18 mcg Inhalation Powder once daily free combination treatment in patients with stable moderate to severe COPD.

Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.

DETAILED DESCRIPTION:
The overall objective is to asses the bronchodilator effect of Tiotropium/Salmeterol/Fluticasone combination delivered via Discair® twice daily as compared with original products Seretide Diskus 500 mcg Inhalation Powder twice daily and Spiriva 18 mcg Inhalation Powder once daily free combination treatment in patients with stable moderate to severe COPD.

For formerly diagnosed patients who met all the inclusion criteria and receiving COPD treatment, the day of the screening visit will be based on the completion of a run-in period, with the length determined by the specific medication. During the run-in period, salbutamol (100 μg inhaler) will be prescribed as a rescue medication.

Patients (following run-in period for formerly diagnosed patients) will be randomly assigned to receive Tiotropium/Salmeterol/Fluticasone fixed dose combination as dry powder inhalation delivered via Discair® twice daily or Seretide Diskus 500 mcg Inhalation Powder twice daily and Spiriva 18 mcg Inhalation Powder once daily free combination for 2-days treatment period.

Patients will be evaluated at 4 consecutive visits: baseline (enrollment), screening, treatment and after treatment.

Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥40 years with COPD diagnosis according to the GOLD (The Global Initiative for Chronic Obstructive Lung Disease) strategy.
* Patients who have symptomatic stable moderate to severe COPD diagnosis with post-bronchodilator FEV1/FVC ratio <0.70, and FEV1 <80% of predicted normal value at screening visit.
* Patients with a mMRC score ≥2
* Current smokers or ex-smokers with a smoking history of at least 10 pack-years
* Patients who have an exacerbation within least a year and no exacerbation within last 4 weeks
* Females patients with childbearing potential using effective birth control method
* Patients who has a capability of communicate with investigator
* Patients who accept to comply with the requirements of the protocol
* Patients who signed written informed consent prior to participation

Exclusion Criteria:

* History of hypersensitivity to drugs contains long acting beta-2 agonists, corticosteroids, anticholinergics or lactose.
* History of asthma or significant chronic respiratory diseases except COPD.
* Patients who had COPD exacerbation or lower respiratory track infections that required antibiotic, oral or parenteral corticosteroid treatment within 4 weeks prior to screening visit or during run-in period.
* Patients with serum potassium level ≤ 3.5 mEq/L or >5.5 mEq/L
* Patients who used systemic corticosteroids or immunosupresants within 4 weeks prior to study onset
* Patients who have a history of myocardial infarction, hearth failure, acute ischemic coroner disease or severe cardiac arrhythmia requiring treatment within least 6 weeks
* Patients who have lung cancer
* Patients who had lung volume reduction operation
* Patients who had live attenuated vaccines within 2 weeks prior to screening visit or during run-in period
* Women patients who are pregnant or nursing
* History of allergic rhinitis or atopy
* Known symptomatic prostatic hypertrophy requiring drug therapy or operation

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Mean max change (ml) from baseline in FEV1 over a period of 48 hrs. | 48 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
Mean % change from baseline in FEV1 over a period of 48 hrs. | 48 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
Mean max change (ml) from baseline in FVC over a period of 48 hrs. | 48 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
Mean % change from baseline in FVC over a period of 48 hrs. | 48 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
FEV1 (AUC0-12) response [AUC: area under the curve; response defined as change from baseline] | Day 1: 0-12 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
FVC (AUC0-12) response | Day 1: 0-12 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
FEV1 (AUC12-24) response | Day 1: 12-24 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
FVC (AUC12-24) response | Day 1: 12-24 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
FEV1 (AUC24-48) response | Day 2: 0-24 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
FVC (AUC24-48) response | Day 2: 0-24 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
FEV1 (AUC0-48) response | 48 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
FVC (AUC0-48) response | 48 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.

SECONDARY OUTCOMES:
The time to onset of bronchodilator effect | 48 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
The time to onset of maximum effect | 48 hrs
  Spirometric measurements will be performed totally at 15 different time points at pretreatment and post-treatment (pre-dose, 15. min, 30. min, 1. hr, 2. hr, 4.hr, 8.hr and 12.hr) during the first treatment day and at 16 different time points (15. min, 30. min, 1. hr, 2. hr, 4.hr, 6 hr, 8.hr and 12.hr) during the second treatment day.
Evaluation of safety of study drug | 48 hrs
  Number of participants with treatment-related adverse events and/or abnormal laboratory values.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Cukurova University Faculty of Medicine, Chest Diseases Department, Adana
  - Health Sciences University, Sureyyapasa Chest Diseases and Thoracic Surgery Training and Research Hospital, Istanbul